CLINICAL TRIAL: NCT05137249
Title: The Glycocalyx in COVID-19 Patients. A Pilot Study
Acronym: Glycovid-19
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Judith Schiefer, Principal Investigator, Medical University of Vienna
Other Study IDs: EK Nr: 1590/2020
Record Dates: First submitted 2021-11-24; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: COVID-19; Endothelial Dysfunction; Coagulation Disorder
Keywords: glycocalyx, covid-19, ards, icu, coagulation,
MeSH Terms: conditions — COVID-19; Hemostatic Disorders; Acute Lung Injury; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with COVID 19 disease: Patients diagnosed with and hospitalized due to COVID-19. Subgroups: ICU admitted COVID-19 + patients vs COVID 19 pts. at normal ward-
- Healthy volunteers: healthy volnuteers

SUMMARY:
The damage of the endothelial glycocalyx is based on microvascular endothelial dysfunction and typical for critical clinical conditions like sepsis, trauma, bleeding, shock, as well as ARDS. We aim to generate first hints regarding the impact of covid-19 disease on the (damage) of the endothelial glycocalyx. Furthermore, we want to investigate the potential coagulopathies, which go along with shedding of the glycocalyx. The detection of and the relation between the severity of the disease, as well as the extent of the glycocalyx damage during the observational period, as well as the hemostatic alterations, are aim of the study.

DETAILED DESCRIPTION:
The damage of the endothelial glycocalyx is based on microvascular endothelial dysfunction and typical for critical clinical conditions like sepsis, trauma, bleeding, shock, as well as ARDS. We aim to generate first hints regarding the impact of covid-19 disease on the (damage) of the endothelial glycocalyx. Furthermore, we want to investigate the potential coagulopathies, which go along with shedding of the glycocalyx. The detection of and the relation between the severity of the disease, as well as the extent of the glycocalyx damage during the observational period, as well as the hemostatic alterations, are aim of the study.Circulating plasma syndecan-1 is measured as surrogat parameter for the extent of the glycocalyx damage.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 detected by PCR measures going along with clinical symptoms
* age > 18 years

Exclusion Criteria:

* refusal of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed and hospitalized with COVID 19 due to clinical symptoms.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
extent of endothelial damage | up to 2 months
  circulating plasma syndecan-1 as surrogat parameter for endothelial damage is measures

CONTACTS AND LOCATIONS:
Overall Officials: Judith Schiefer, MD PhD, Principal Investigator — Medical University of Vienna, Department of Anesthesia, Intensive Care Medicine and Pain Medicine
Locations (1):
- Medical University of Vienna, Vienna, Austria